CLINICAL TRIAL: NCT03429673
Title: A Multi-centre Real-world Non-interventional Observational Study to Evaluate Effectiveness and Safety of Surgeries in the Chinese Early-stage Patients With Non-small Cell Lung Cancer
Brief Title: A Study to Evaluate Effectiveness and Safety of Surgeries in Elderly NSCLC Patients
Status: Completed | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Deruo Liu, Professor, China-Japan Friendship Hospital
Other Study IDs: CJ-LC-01
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Chinese; real-world evidences; NSCLC; surgeries
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with surgeries: Pathologically diagnosed elderly early Chinese patients with non-small cell lung cancer who received lobectomy or segment/wedge dissection
  Interventions: Procedure: Surgeries

INTERVENTIONS:
Procedure: Surgeries — Lobectomy or segment/wedge dissection

SUMMARY:
The trial was designed to compare effectiveness and safety of surgeries in the patients with non-small cell lung cancer

DETAILED DESCRIPTION:
The trial is a multi-centre, real-world, non-interventional, observational study. The Chinese elderly pathologically diagnosed patients with early-stage non-small cell lung cancer enrolled from 2015 to 2017 who received lobectomy or segment/wedge dissection were included and the study data on patient demographic/tumor biological characteristics, and clinical treatments were retrospectively collected to evaluate effectiveness and safety of the surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received surgeries from 2014 to 2017;
* Patients who received lobectomy or segment/wedge dissection;
* Pathologically diagnosed patients with non-small cell lung cancer;
* Patients with age >=65 years old.

Exclusion Criteria:

* Patients who received neoadjuvant therapy prior to surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Pathological diagnosed elderly Chinese patients with non-small cell lung cancer who received lobectomy or segment/wedge dissection
Sampling Method: Non-Probability Sample
Enrollment: 10885 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2015-2017
  Overall survival

OTHER OUTCOMES:
Overall survivals in the subgroups | 2015-2017
  Overall survivals in the subgroups categorised by age, tumor size, and clinical/pathological staging
Impact factors of overall survival | 2015-2017
  Impact factors of overall survival as measured by patient demographic/tumor biological characteristics
Death rate within 30/90 days after surgeries | 2015-2017
  Death rate within 30/90 days after surgeries
Incidence of perioperative complications | 2015-2017
  Incidence of perioperative complications

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China People's Liberation Army Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huaxi Technology University, Wuhan, Hubei
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliate to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Feng H, Zhao H, Hu J, Liu L, Liu Y, Li X, Xu L, Li Y, Lu X, Fu X, Yang H, Liu D. Sublobar resection is associated with better perioperative outcomes in elderly patients with clinical stage I non-small cell lung cancer: a multicenter retrospective cohort study. J Thorac Dis. 2019 May;11(5):1838-1848. doi: 10.21037/jtd.2019.05.20. PMID 31285876